CLINICAL TRIAL: NCT05180955
Title: The Role of Clamping Before Removal of a Pneumothorax Drain Connected to a Digital Drainage System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Wytze de Boer, MD, Isala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Chest Tube Removal 001
Record Dates: First submitted 2021-12-07; First posted 2022-01-06 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Pneumothorax and Air Leak
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: The study will be conducted as a, prospective, open label, non-inferiority, randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital drainage system group (Other): chest tube removal will be determined by air flow criteria as indicated by the digital drainage system data.
  Interventions: Other: Digital drainage system
- Digital drainage system + clamping trial group (Other): In the control group removal will be determined by the same criteria of the digital drainage system but before removal, a chest tube clamping test will be performed.
  Interventions: Other: Digital drainage system + clamping trial

INTERVENTIONS:
Other: Digital drainage system — In the intervention group; chest tube removal will be determined by air flow criteria as indicated by the digital drainage system data, the tube will not be clamped.
  Arms: Digital drainage system group
Other: Digital drainage system + clamping trial — In the control group removal will be determined by the same criteria of the digital drainage system but before removal, a chest tube clamping test will be performed.
  Arms: Digital drainage system + clamping trial group

SUMMARY:
The study will be conducted as a, prospective, open label, non-inferiority, randomized controlled trial. In the intervention group; chest tube removal will be determined by air flow criteria as indicated by the digital drainage system data. In the control group removal will be determined by the same criteria of the digital drainage system but before removal, a chest tube clamping test will be performed. Primary outcome measure: recurrent pneumothorax after chest tube removal requiring chest tube reinsertion

DETAILED DESCRIPTION:
Determining and timing of chest tube removal has been a continuous topic of debate amongst both surgeons and pulmonologist. It is plausible that provocative clamping tests are no longer necessary when a digital continuous recording drainage device is used that demonstrates the absence of (intermittent) air leak. However, clamping trials are still performed in clinical care, it is an expert opinion's policy prompted by fear of recurrent pneumothorax and no comparative studies exist. We hypothesize that chest tube removal exclusively based on digital drainage system data is as safe as adding a clamping test before removal in patients treated for pneumothorax or after lung surgery.

The study will be conducted as a, prospective, open label, non-inferiority, randomized controlled trial. In the intervention group; chest tube removal will be determined by air flow criteria as indicated by the digital drainage system data. In the control group removal will be determined by the same criteria of the digital drainage system but before removal, a chest tube clamping test will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Digital chest tube drainage system
* Pneumothorax (primary, secondary, pulmonary surgery)

Exclusion Criteria:

* Pleural effusion as primary indication for chest tube placement.
* Empyema
* Suspected chest tube malfunction (e.g., leaking, occlusion, malposition)
* Intubated during chest tube removal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Recurrent pneumothorax after chest tube removal | 0-24 hours after drain removal
  number of patients requiring chest tube reinsertion within 24 hours after chest tube removal for recurrent pneumothorax

CONTACTS AND LOCATIONS:
Overall Officials: Jos Stigt, MD PhD, Study Director — Isala
Locations (1):
- Isala Klinieken, Zwolle, Overijssel, Netherlands

IPD SHARING:
Plan to Share IPD: No